CLINICAL TRIAL: NCT04424862
Title: Multitarget Therapy for Idiopathic Membranous Nephropathy
Acronym: MTIMN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wenhu Liu, Director, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 3 20200607
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Efficacy
MeSH Terms: interventions — Prednisone; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multitarget Therapy (Experimental): The combined therapy with prednisone, ciclosporin and mycophenolate mofetil.
  Interventions: Drug: Prednisone, ciclosporin and mycophenolate mofetil
- Control (Active Comparator): Ponticelli Regimen
  Interventions: Drug: Ponticelli Regimen

INTERVENTIONS:
Drug: Prednisone, ciclosporin and mycophenolate mofetil — Multitarget Therapy
  Arms: Multitarget Therapy
Drug: Ponticelli Regimen — Month 1: i.v. methylprednisolone (0.5 g) daily for three doses, then oral prednison (0.5 mg/kg/d, maximum dose 30mg/d) for 27 days Month 2: Oral cyclophosphamide (2.0 mg/kg/d, maximum dose 100mg/d) for 30 days Month 3: Repeat Month 1 Month 4: Repeat Month 2 Month 5: Repeat Month 1 Month 6: Repeat Month 2
  Arms: Control

SUMMARY:
Membranous nephropathy (MN) is one of the commonest causes of nephrotic syndrome in adults, idiopathic membranous nephropathy (IMN) accounts for 70%-80% of all MN patients. There is no standard specific treatment for IMN. Initial therapy should be supportive and involves restricting dietary protein and sodium intake, controlling blood pressure, hyperlipidemia, and edema. The best proven therapy for patients with IMN is combined use of corticosteroids and cyclophosphamide. However, there are some potential risk of other serious side effects associated with the use of cytotoxic agents, such as bone marrow toxicity, severe infections, gonadal dysfunction, and the long-term risk of malignancy.

The ideal maintenance treatment scheme for patients with IMN requires not only a remission of nephrotic syndrome but also, fewer adverse effects. Some retrospective study suggested that multitarget therapy (prednisone+calcineurin inhibitors+mycophenolate mofetil) was effective for refractory IMN. However, we cannot get confirmed conclusion from the previous study due to the limitation of retrospective studies with small sample size.

In this prospective multicenter randomized trial, we compared the efficacy between multitarget therapy and Ponticelli regimen.

Trial Aims and Hypothesis The specific aims of this trial are to test the hypothesis

1. that multitarget therapy is non-inferior to Ponticelli regimen in inducing long-term remission (CR or PR) of proteinuria in patients with IMN.
2. that multitarget therapy reduces the number of relapses (efficacy in sustaining remission) and increases the time to relapse when compared with treatment with Ponticelli regimen.
3. that multitarget therapy has a better side-effect profile when compared with treatment with Ponticelli regimen in patients with IMN.

Methods:

Patient Recruitment Inclusion and exclusion criteria are as follows.

Inclusion Criteria:

* Age: 18-70 years.
* Body weight: 50-90 kg.
* Patients with membranous nephropathy were eligible if their diagnosis was confirmed by renal biopsy, with the biopsy sample examined by light, immunofluorescence, and electron microscopy. Renal biopsy samples were reviewed by the two principal investigators and two renal pathologists.
* IMN patients with moderate risk and have a decline of less than 50% in proteinuria despite renin-angiotensin system blockade for at least 6 months before randomization. OR, IMN patients with high risk or very high risk.
* Serum albumin < 30 g/L.
* eGFR by MDRD formula had to be ≥ 60 ml/min per 1.73 m2.

Exclusion criteria:

* Secondary MN, pregnancy, breastfeeding, immunosuppressive treatment in the 3 preceding months, and active infectious disease.
* Hepatitis B serology included Hbs antigen and Hbs and Hbc antibodies. Patients with active hepatitis B and those with past hepatitis B infection without anti-Hbs antibodies will be excluded.
* Patients with reproductive demand will be excluded.

Randomization and Treatment Groups Once all entry criteria have been satisfied and confirmed, patients will be randomized to treatment with multitarget therapy or Ponticelli regimen.

Multitarget therapy:

Combination with prednisone, ciclosporin and mycophenolate mofetil.

Ponticelli regimen:

Cyclical corticosteroid/alkylating-agent therapy for IMN. Outcomes Primary outcome: The primary clinical outcome was the composite of complete or partial remission at 12 months.

Secondary outcome: the composite of complete or partial remission at 6 months; complete remission at 6 months; and adverse events, relapse.

DETAILED DESCRIPTION:
Membranous nephropathy (MN) is one of the commonest causes of nephrotic syndrome in adults, idiopathic membranous nephropathy (IMN) accounts for 70%-80% of all MN patients. There is no standard specific treatment for IMN. Initial therapy should be supportive and involves restricting dietary protein and sodium intake, controlling blood pressure, hyperlipidemia, and edema. The best proven therapy for patients with IMN is combined use of corticosteroids and cyclophosphamide. However, there are some potential risk of other serious side effects associated with the use of cytotoxic agents, such as bone marrow toxicity, severe infections, gonadal dysfunction, and the long-term risk of malignancy.

The ideal maintenance treatment scheme for patients with IMN requires not only a remission of nephrotic syndrome but also, fewer adverse effects. Some retrospective study suggested that multitarget therapy (prednisone+calcineurin inhibitors+mycophenolate mofetil) was effective for refractory IMN. However, we cannot get confirmed conclusion from the previous study due to the limitation of retrospective studies with small sample size.

In this prospective multicenter randomized trial, we compared the efficacy between multitarget therapy and Ponticelli regimen.

Trial Aims and Hypothesis The specific aims of this trial are to test the hypothesis

1. that multitarget therapy is non-inferior to Ponticelli regimen in inducing long-term remission (CR or PR) of proteinuria in patients with IMN.
2. that multitarget therapy reduces the number of relapses (efficacy in sustaining remission) and increases the time to relapse when compared with treatment with Ponticelli regimen.
3. that multitarget therapy has a better side-effect profile when compared with treatment with Ponticelli regimen in patients with IMN.

Methods:

Patient Recruitment Inclusion and exclusion criteria are as follows.

Inclusion Criteria:

* Age: 18-70 years.
* Body weight: 50-90 kg.
* Patients with membranous nephropathy were eligible if their diagnosis was confirmed by renal biopsy, with the biopsy sample examined by light, immunofluorescence, and electron microscopy. Renal biopsy samples were reviewed by the two principal investigators and two renal pathologists.
* IMN patients with moderate risk and have a decline of less than 50% in proteinuria despite renin-angiotensin system blockade for at least 6 months before randomization. OR, IMN patients with high risk or very high risk.
* Serum albumin < 30 g/L.
* eGFR by MDRD formula had to be ≥ 60 ml/min per 1.73 m2.

Exclusion criteria:

* Secondary MN, pregnancy, breastfeeding, immunosuppressive treatment in the 3 preceding months, and active infectious disease.
* Hepatitis B serology included Hbs antigen and Hbs and Hbc antibodies. Patients with active hepatitis B and those with past hepatitis B infection without anti-Hbs antibodies will be excluded.
* Patients with reproductive demand will be excluded.

Randomization and Treatment Groups Once all entry criteria have been satisfied and confirmed, patients will be randomized to treatment with multitarget therapy or Ponticelli regimen.

Multitarget therapy:

The patients in the multitarget group continued to receive prednisone 1 mg/kg/d (maximum dosage 60mg/d) for 2 weeks and then tapered by 5mg per week. When reduced to 30mg/d, maintained for 1 month, and then tapered by 5 mg per month. When reduced to 20mg/d, maintained for 2 months, and then tapered by 2.5 mg per two-month. When reduced to 5 mg/d, maintained for 4 months.

Mycophenolate mofetil (1 g/d for 6 months and then tapered to 0.75 g/d for another 12 months, and tapered 0.5g for another 12 months) Ciclosporin (initial dosage 100 mg/d, and adjusted the dosage to maintain trough concentration at 80-120 ng/mL. If the patients get complete remission during dosage adjustment period, then maintain the dosage, don't need to get to the target trough concentration. (1) When the patients get complete remission, maintain the dosage for 2 weeks, then tapered by 25mg/d per 3 months. When reduced to 50 mg/d, maintain for 12 months, then tapered to 25mg/d for another 12 months. (2) When the patients only get partial remission, maintain the target dosage for 12 months, and then adjust the dosage followed "(1)". (3) When the patients no response, maintain the target dosage for 6 months, if the decreased UTP < 25%, suggested change the therapy regimen. If the decreased UTP ≥ 25%, maintain the dosage for another 6 months, then follow "(2)".

Ponticelli regimen:

Cyclical corticosteroid/alkylating-agent therapy for IMN. Outcomes Primary outcome: The primary clinical outcome was the composite of complete or partial remission at 12 months.

Secondary outcome: the composite of complete or partial remission at 6 months; complete remission at 6 months; and adverse events, relapse.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years.
* Body weight: 50-90 kg.
* Patients with membranous nephropathy were eligible if their diagnosis was confirmed by renal biopsy, with the biopsy sample examined by light, immunofluorescence, and electron microscopy. Renal biopsy samples were reviewed by the two principal investigators and two renal pathologists.
* IMN patients with moderate risk and have a decline of less than 50% in proteinuria despite renin-angiotensin system blockade for at least 6 months before randomization. OR, IMN patients with high risk or very high risk.
* Serum albumin < 30 g/L.
* eGFR by MDRD formula had to be ≥ 60 ml/min per 1.73 m2.

Exclusion criteria:

* Secondary MN, pregnancy, breastfeeding, immunosuppressive treatment in the 3 preceding months, and active infectious disease.
* Hepatitis B serology included Hbs antigen and Hbs and Hbc antibodies. Patients with active hepatitis B and those with past hepatitis B infection without anti-Hbs antibodies will be excluded.
* Patients with reproductive demand will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
The composite of complete or partial remission at 12 months | Month 12
  complete remission: proteinuria of no more than 0.3 g per 24 hours and a serum albumin level of at least 35 g per milliliter. Partial remission: a reduction in proteinuria of at least 50% from baseline plus final proteinuria between 0.3 g and 3.5 g per 24 hours regardless of creatinine clearance or the serum albumin level.

SECONDARY OUTCOMES:
Composite of complete or partial remission at 6 months | at momth 6
  complete remission: proteinuria of no more than 0.3 g per 24 hours and a serum albumin level of at least 35 g per milliliter. Partial remission: a reduction in proteinuria of at least 50% from baseline plus final proteinuria between 0.3 g and 3.5 g per 24 hours regardless of creatinine clearance or the serum albumin level.
Treatment failure | at momth 6
  proteinuria decreased no more than 25% of baseline at month
adverse events | within 12 months
  Advers events happened during study period
Relapse | within 12 months
  Relapse during study period

CONTACTS AND LOCATIONS:
Overall Officials: Zongli Diao, MD, Principal Investigator — Beijing Frienship Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Frienship Hospital, Capital Medical University, Beijing, Beijing Municipality